CLINICAL TRIAL: NCT03428490
Title: Developing and Evaluating a Fully Integrated Treatment Program for Comorbid Social Anxiety and Alcohol Use Disorders
Brief Title: Treatment for Comorbid Social Anxiety and Alcohol Use Disorders.
Acronym: FIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Matrix Institute on Addictions (Unknown)
Responsible Party: Principal Investigator, Kate Taylor, Assistant Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SOCANX1; 1R34AA025364-01 (NIH)
Record Dates: First submitted 2017-11-16; First posted 2018-02-09 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Alcohol Use Disorder; Social Anxiety Disorder
Keywords: Integrated Treatment; Alcohol Use Disorder; Social Anxiety Disorder; Comorbidity; Cognitive Behavioral Therapy
MeSH Terms: conditions — Alcoholism; Phobia, Social

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomized to the Fully Integrated Treatment (FIT; N =30) or usual care in the Matrix Institute IOP (UC; N = 30).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fully Integrated Treatment (Experimental): Evidence-based substance use treatment combined with Cognitive Behavioral Therapy (CBT) for Social Anxiety Disorder Intervention name: Fully integrated treatment
  Interventions: Behavioral: Fully integrated treatment
- Usual Intensive Outpatient Care (Active Comparator): Evidence-based substance use disorder treatment Intervention name: Stand-alone Intensive Outpatient Program
  Interventions: Behavioral: Stand-alone Intensive Outpatient Program

INTERVENTIONS:
Behavioral: Fully integrated treatment — Clinicians will be delivering CBT for Social Anxiety Disorder directly into the context of the Matrix's evidence-based treatment for substance use disorders (i.e., The Matrix Model).
  Arms: Fully Integrated Treatment
Behavioral: Stand-alone Intensive Outpatient Program — Evidence-based treatment for substance use disorders (i.e., The Matrix Model).
  Arms: Usual Intensive Outpatient Care

SUMMARY:
Alcohol use disorders (AUD) and social anxiety disorder (SAD) are highly comorbid and associated with significant impairment. Social anxiety comorbidity is associated with poorer addiction treatment engagement and outcomes. Thus, addressing underlying SAD symptoms that may lead to and maintain alcohol problems, as well as undermine successful treatment for AUD, is warranted. This proposal aims to develop and evaluate a fully integrated outpatient program for comorbid SAD and AUD that weaves evidence-based treatment for SAD (i.e., exposure-based cognitive behavioral therapy) into a traditional, evidence-based treatment for AUD.

First, the investigators will develop the protocol for the fully integrated treatment (FIT). The overarching goal of FIT will be to simultaneously deliver AUD and SAD treatment. Development will be an iterative process guided by previous research (including our own), and by input from clinicians, administrators, and patients in an outpatient substance use disorder treatment clinic. After the protocol is developed, the investigators will use their established clinician training procedures to train clinicians at their community partnered clinic to competently deliver the intervention. After protocol development and clinician training, the investigators will conduct a pilot randomized clinical trial (RCT) comparing the efficacy of our fully integrated treatment (FIT) for comorbid alcohol use and social anxiety disorders to usual care (UC) in the community substance use disorder specialty clinic. The goals of the RCT will be to gather data regarding acceptability, feasibility, and preliminary efficacy of the FIT protocol. The investigators will randomize treatment-seeking participants (N = 60) who have comorbid SAD and AUD. The investigators will assess treatment engagement, social anxiety outcomes, and alcohol use outcomes at baseline, 3-months, and 6-months from baseline. The investigators will also gather qualitative and quantitative acceptability data from patients after completing FIT, which may guide final refinements of FIT prior to testing in a larger-scale grant.

The knowledge gained from this investigation has the potential to significantly improve the treatment of alcohol use disorders and make a significant public health impact. The focus on direct translation to community practice paradigms and the emphasis on full mental health and addiction treatment integration significantly advance the field.

DETAILED DESCRIPTION:
In this study, potential participants will be screened either by University of California, Los Angeles (UCLA) staff or at the Matrix Institute on Addiction to determine whether they may have social anxiety and alcohol use disorder symptoms. If they screen positive for these symptoms, they will be invited to come in for a comprehensive baseline assessment consisting of interviews, questionnaires, and a behavioral assessment. Eligible participants will be randomly assigned to either receive standard Matrix treatment consisting of a 9-hour per week Intensive Outpatient Program (IOP) lasting approximate 2-3 months; or FIT, an Intensive Outpatient Program (also 9 hours per week for approximately 2-3 months) consisting of cognitive behavioral therapy (CBT) for social anxiety disorder that is woven into the alcohol recovery program. After treatment, participants will complete another assessment, and then will complete one several months later.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be currently enrolled in the IOP at Matrix Institute (our community partner) for the treatment of their alcohol use disorder;
* fluent in English;
* meet the DSM-5 criteria for social anxiety disorder and alcohol use disorder

Exclusion Criteria:

* marked cognitive impairment
* moderate to severe suicidality
* unstable manic or psychotic symptoms.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Alcohol consumption at 3 and 6 months | Baseline, 3 months, and 6 months
  The Timeline Followback (TLFB), a gold standard semi-structured interview measure of alcohol consumption, will be used in order to obtain number of drinking days
Change from Baseline Social Anxiety Symptoms in Situations at 3 and 6 months | Baseline, 3 months, and 6 months
  The Leibowitz Social Anxiety Scale-Self Report (LSAS-SR) will be used to assess the extent to which individuals are anxious in, and avoid, a variety of social situations, including performance based and social-interactional situations. Anxiety and avoidance are each rated from 1 (none/never) to 4 (extreme/always) Higher scores indicate greater severity of social anxiety.

SECONDARY OUTCOMES:
Change from Baseline Social anxiety-related drinking motives at 3 and 6 months | Baseline, 3 months, and 6 months
  This will be assessed using the Drinking to Cope with Social Anxiety Scale (DCSAS), which measures drinking behavior in social situations. The score on the measure is out of 72, with a minimum score of 0 indicating the least amount of avoidance/drinking to scope in situations, and 72 indicating the most amount of avoidance/drinking to scope in situations
Change from Baseline Quality of Life and overall functioning at 3 and 6 months | Baseline, 3 months, and 6 months
  This will be assessed using the Short Form (SF-8), which is a generic quality of life measure with 8 items. The total score is out of 41, with a minimum score of 8 indicating best quality of life score and a maximum score or 41 indicating worst quality of life score.
Change from Baseline Alcohol Problems at 3 and 6 months | Baseline, 3 months, and 6 months
  The Short Inventory of Problems, a dimensional measure of alcohol-related consequences, will be used using "past month" as the time frame for each assessment.
Change from Baseline Alcohol Drinks per Day at 3 and 6 months | Baseline, 3 months, and 6 months
  The Timeline Followback (TLFB) will be used in order to obtain average drinks per drinking day
Change from Baseline Heavy Alcohol Use Days at 3 and 6 months | Baseline, 3 months, and 6 months
  The Timeline Followback (TLFB) will be used in order to obtain % of heavy drinking days (defined as ≥4 drinks per day for women and ≥5 drinks per day for men)
Change from Baseline Alcohol Abstinence at 3 and 6 months | Baseline, 3 months, and 6 months
  The Timeline Followback (TLFB) will be used in order to obtain sustained abstinence (v. not) during the past 30 days
Change from Baseline Social Anxiety Symptom Severity at 3 and 6 months | Baseline, 3 months, and 6 months
  The Behavioral Approach Task (BAT), a validated behavioral assessment of social anxiety severity, will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Kate Wolitzky-Taylor, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Matrix Institute on Addictions, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No